CLINICAL TRIAL: NCT04795089
Title: Gait Pattern, Experienced Global Change, Sense of Coherence, Quality of Life, Anxiety and Depression Symptoms After Shunt Surgery in Idiopathic Normal Pressure Hydrocephalus, in Relation With Healthy Individuals
Brief Title: Gait Pattern and Experienced Global Change After Shunt Surgery in Idiopathic Normal Pressure Hydrocephalus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Fredrik Lundin, Principal Investigator, Linkoeping University
Other Study IDs: 2020-00719
Record Dates: First submitted 2021-02-18; First posted 2021-03-12 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Idiopathic Normal Pressure Hydrocephalus
Keywords: gait analysis; outcome; surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with iNPH and shunt surgery.
  Interventions: Procedure: Shunt surgery
- Healthy individuals: Healthy controls with similar gender and age distribution as the patients.

INTERVENTIONS:
Procedure: Shunt surgery — Patients are evaluated before and after shunt surgery which is a standard intervention in the clinical practice. HI do not undergo intervention.
  Groups: Patients

SUMMARY:
Part 1 Patients with idiopathic Normal Pressure Hydrocephalus (iNPH) have variable disabilities regarding gait, balance, cognition and continence. Analysis of the gait pattern in iNPH has an important part in clinical diagnosing and evaluation of outcome after shunt surgery. The gait pattern is only partly explained and more detailed information about gait in iNPH is needed in relation with ordinary clinical measurements.

Part 2 Approximately 70 % of patients with iNPH improve after shunt surgery. Commonly different grading scales and measurements regarding functions are used in the evaluation. To some extent, patients improve in Quality of life after surgery (QoL). In this study, the patient´s own grading of improvements in relation with QoL, sense of coherence (SOC) and symptoms of depression and anxiety are analyzed.

DETAILED DESCRIPTION:
Consecutive patients with iNPH, which are planed for shunt surgery at the neurological and neurosurgical departments of University Hospital of Linköping, are included. Before operation and 3 months postoperatively, the patient´s gait pattern are analyzed with RehaGait analysis system. The patients also fill in a questionnaire about SOC, QoL and symptoms of depression and anxiety at these assessment sessions. Additionally at the follow up, the patients are grading their overall experienced change and specified changes in gait, balance, continence and neuropsychology with the global Rating of Change Scale (GRC-scale). At baseline and at follow up, the patients also perform the ordinary clinical assessments with measurements covering the domains gait, balance, continence and neuropsychology in the iNPH-scale. A convenience sample of Healthy individuals aged > 60 years, conduct the same questionnaires: SOC, QoL and symptoms of depression and anxiety and perform the RehaGait analysis system once.

ELIGIBILITY:
Inclusion criteria for patients:

* iNPH-diagnosis according to the international guidelines (2005)
* Planed for shunt surgery

Exclusion criteria for patients:

* Cognitive impairment that makes it impossible to participate
* Not able to walk 20 meters without walking aids (part 1)

Inclusion criteria for healthy individuals:

* > 60 years of age
* Subjectively healthy without any serious disease

Exclusion criteria healthy individuals:

* Visible gait- or balance disturbance
* Dementia diagnosis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients: Al consecutively available patients evaluated for iNPH at Neurology department Linköping University hospital.
  HI: Convenience sample among relatives, friends and using advertising.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Gait pattern assessed with the Hasomed RehaGait analyzer pro. Variable: Analyzed steps (number). | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 1. Mobile gait analysis system.
Gait pattern assessed with the Hasomed RehaGait analyzer pro. Variable: Analyzed distance (m) | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 1. Mobile gait analysis system.
Gait pattern assessed with the Hasomed RehaGait analyzer pro. Variable: Stride duration (seconds) | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 1. Mobile gait analysis system.
Gait pattern assessed with the Hasomed RehaGait analyzer pro. Variable: Stride length (cm) | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 1. Mobile gait analysis system.
Gait pattern assessed with the Hasomed RehaGait analyzer pro. Variable: Cadence (steps per minute) | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 1. Mobile gait analysis system.
Gait pattern assessed with the Hasomed RehaGait analyzer pro. Variable: Gait phases (seconds) | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 1. Mobile gait analysis system.
Gait pattern assessed with the Hasomed RehaGait analyzer pro. Variable: Heel strike and Toe of angle (angle degree) | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 1. Mobile gait analysis system.
Gait pattern assessed with the Hasomed RehaGait analyzer pro. Variable: Circumduction (cm) | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 1. Mobile gait analysis system.
Gait pattern assessed with the Hasomed RehaGait analyzer pro. Variable: Ankle joint angle (degree of angle) | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 1. Mobile gait analysis system.
Gait pattern assessed with the Hasomed RehaGait analyzer pro. Variable: Knee joint angle (degree of angle) | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 1. Mobile gait analysis system.
Gait pattern assessed with the Hasomed RehaGait analyzer pro. Variable:Hip joint angle (degree of angle) | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 1. Mobile gait analysis system.
Grading of severity in idiopathic normal pressure hydrocephalus assessed with the Idiopathic Normal Pressure Hydrocephalus Scale | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 1 and part 2. Scores 0-100, higher scores mean a better outcome.
Mobility, walking ability and balance assessed with the Timed up and Go test | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 1. Variables: Time in seconds and number of steps.
Rating of global change assessed with the Global Rating of Change Scale | Rating at 3 month follow-up for patients.
  Measurement in part 2. Scores -5-5 in global change, gait, balance, continence and cognition. Higher scores mean a better outcome.
Sense of Coherence assessed with the 29 item Orientation to life questionnaire - swedish version (KASAM questionnaire) | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 2. Scores 29-203, higher scores mean a better outcome.
Anxiety and depression assessed with the Hospital Anxiety and Depression Scale | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 2. Anxiety scores 0-21, Depression scores 0-21, lower scores mean a better outcome.
Health-related quality of life assessed with EQ-5D-5L | Change from baseline to 3 month follow-up for patients. Once for HI.
  Measurement in part 2. Scores 5-25, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Lundin, PhD, Study Director — Neurology department, Linköping University Hospital
Locations (1):
- Neurology department, Linköping University Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Relkin N, Marmarou A, Klinge P, Bergsneider M, Black PM. Diagnosing idiopathic normal-pressure hydrocephalus. Neurosurgery. 2005 Sep;57(3 Suppl):S4-16; discussion ii-v. doi: 10.1227/01.neu.0000168185.29659.c5. PMID 16160425
- [Background] Klinge P, Hellstrom P, Tans J, Wikkelso C; European iNPH Multicentre Study Group. One-year outcome in the European multicentre study on iNPH. Acta Neurol Scand. 2012 Sep;126(3):145-53. doi: 10.1111/j.1600-0404.2012.01676.x. Epub 2012 May 10. PMID 22571428
- [Background] Shore WS, deLateur BJ, Kuhlemeier KV, Imteyaz H, Rose G, Williams MA. A comparison of gait assessment methods: Tinetti and GAITRite electronic walkway. J Am Geriatr Soc. 2005 Nov;53(11):2044-5. doi: 10.1111/j.1532-5415.2005.00479_9.x. No abstract available. PMID 16274403
- [Background] Schniepp R, Trabold R, Romagna A, Akrami F, Hesselbarth K, Wuehr M, Peraud A, Brandt T, Dieterich M, Jahn K. Walking assessment after lumbar puncture in normal-pressure hydrocephalus: a delayed improvement over 3 days. J Neurosurg. 2017 Jan;126(1):148-157. doi: 10.3171/2015.12.JNS151663. Epub 2016 Mar 18. PMID 26991388
- [Background] Selge C, Schoeberl F, Zwergal A, Nuebling G, Brandt T, Dieterich M, Schniepp R, Jahn K. Gait analysis in PSP and NPH: Dual-task conditions make the difference. Neurology. 2018 Mar 20;90(12):e1021-e1028. doi: 10.1212/WNL.0000000000005168. Epub 2018 Feb 21. PMID 29467306
- [Background] Lim YH, Ko PW, Park KS, Hwang SK, Kim SH, Han J, Yoon U, Lee HW, Kang K. Quantitative Gait Analysis and Cerebrospinal Fluid Tap Test for Idiopathic Normal-pressure Hydrocephalus. Sci Rep. 2019 Nov 7;9(1):16255. doi: 10.1038/s41598-019-52448-3. PMID 31700018
- [Background] Najafi B, Helbostad JL, Moe-Nilssen R, Zijlstra W, Aminian K. Does walking strategy in older people change as a function of walking distance? Gait Posture. 2009 Feb;29(2):261-6. doi: 10.1016/j.gaitpost.2008.09.002. Epub 2008 Oct 25. PMID 18952435
- [Background] Konig N, Singh NB, von Beckerath J, Janke L, Taylor WR. Is gait variability reliable? An assessment of spatio-temporal parameters of gait variability during continuous overground walking. Gait Posture. 2014;39(1):615-7. doi: 10.1016/j.gaitpost.2013.06.014. Epub 2013 Jul 6. PMID 23838361
- [Background] Donath L, Faude O, Lichtenstein E, Pagenstert G, Nuesch C, Mundermann A. Mobile inertial sensor based gait analysis: Validity and reliability of spatiotemporal gait characteristics in healthy seniors. Gait Posture. 2016 Sep;49:371-374. doi: 10.1016/j.gaitpost.2016.07.269. Epub 2016 Jul 30. PMID 27494305
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Hellstrom P, Klinge P, Tans J, Wikkelso C. A new scale for assessment of severity and outcome in iNPH. Acta Neurol Scand. 2012 Oct;126(4):229-37. doi: 10.1111/j.1600-0404.2012.01677.x. Epub 2012 May 16. PMID 22587624
- [Background] Toma AK, Papadopoulos MC, Stapleton S, Kitchen ND, Watkins LD. Systematic review of the outcome of shunt surgery in idiopathic normal-pressure hydrocephalus. Acta Neurochir (Wien). 2013 Oct;155(10):1977-80. doi: 10.1007/s00701-013-1835-5. Epub 2013 Aug 23. PMID 23975646
- [Background] Israelsson H, Eklund A, Malm J. Cerebrospinal Fluid Shunting Improves Long-Term Quality of Life in Idiopathic Normal Pressure Hydrocephalus. Neurosurgery. 2020 Apr 1;86(4):574-582. doi: 10.1093/neuros/nyz297. PMID 31504827
- [Background] Junkkari A, Sintonen H, Nerg O, Koivisto AM, Roine RP, Viinamaki H, Soininen H, Jaaskelainen JE, Leinonen V. Health-related quality of life in patients with idiopathic normal pressure hydrocephalus. Eur J Neurol. 2015 Oct;22(10):1391-9. doi: 10.1111/ene.12755. Epub 2015 Jun 24. PMID 26104064
- [Background] Junkkari A, Hayrinen A, Rauramaa T, Sintonen H, Nerg O, Koivisto AM, Roine RP, Viinamaki H, Soininen H, Luikku A, Jaaskelainen JE, Leinonen V. Health-related quality-of-life outcome in patients with idiopathic normal-pressure hydrocephalus - a 1-year follow-up study. Eur J Neurol. 2017 Jan;24(1):58-66. doi: 10.1111/ene.13130. Epub 2016 Sep 19. PMID 27647684
- [Background] Junkkari A, Roine RP, Luikku A, Rauramaa T, Sintonen H, Nerg O, Koivisto AM, Hayrinen A, Viinamaki H, Soininen H, Jaaskelainen JE, Leinonen V. Why Does the Health-Related Quality of Life in Idiopathic Normal-Pressure Hydrocephalus Fail to Improve Despite the Favorable Clinical Outcome? World Neurosurg. 2017 Dec;108:356-366. doi: 10.1016/j.wneu.2017.08.170. Epub 2017 Sep 5. PMID 28887286
- [Background] Cage TA, Auguste KI, Wrensch M, Wu YW, Gupta N. Self-reported functional outcome after surgical intervention in patients with idiopathic normal pressure hydrocephalus. J Clin Neurosci. 2011 May;18(5):649-54. doi: 10.1016/j.jocn.2010.08.028. Epub 2011 Mar 2. PMID 21371890
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Gallagher R, Marquez J, Osmotherly P. Clinimetric Properties and Minimal Clinically Important Differences for a Battery of Gait, Balance, and Cognitive Examinations for the Tap Test in Idiopathic Normal Pressure Hydrocephalus. Neurosurgery. 2019 Jun 1;84(6):E378-E384. doi: 10.1093/neuros/nyy286. PMID 30010977
- [Background] Langius A, Bjorvell H, Antonovsky A. The sense of coherence concept and its relation to personality traits in Swedish samples. Scand J Caring Sci. 1992;6(3):165-71. doi: 10.1111/j.1471-6712.1992.tb00146.x. PMID 1439378
- [Background] Kristofferzon ML, Engstrom M, Nilsson A. Coping mediates the relationship between sense of coherence and mental quality of life in patients with chronic illness: a cross-sectional study. Qual Life Res. 2018 Jul;27(7):1855-1863. doi: 10.1007/s11136-018-1845-0. Epub 2018 Apr 5. PMID 29623597
- [Background] Sinikallio S, Pakarinen M, Tuomainen I, Airaksinen O, Viinamaki H, Aalto TJ. Preoperative sense of coherence associated with the 10-year outcomes of lumbar spinal stenosis surgery. J Health Psychol. 2019 Jun;24(7):989-997. doi: 10.1177/1359105316687633. Epub 2017 Jan 17. PMID 28810389
- [Background] Israelsson H, Allard P, Eklund A, Malm J. Symptoms of Depression are Common in Patients With Idiopathic Normal Pressure Hydrocephalus: The INPH-CRasH Study. Neurosurgery. 2016 Feb;78(2):161-8. doi: 10.1227/NEU.0000000000001093. PMID 26528670
- [Background] Antonovsky H, Sagy S. The development of a sense of coherence and its impact on responses to stress situations. J Soc Psychol. 1986 Apr;126(2):213-25. No abstract available. PMID 3724090
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Brooks R. EuroQol: the current state of play. Health Policy. 1996 Jul;37(1):53-72. doi: 10.1016/0168-8510(96)00822-6. PMID 10158943
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Derived] Rydja J, Pohl P, Eleftheriou A, Lundin F. Gait characteristics in idiopathic normal pressure hydrocephalus: A controlled study using an inertial sensor system. PLoS One. 2025 Feb 26;20(2):e0317901. doi: 10.1371/journal.pone.0317901. eCollection 2025. PMID 40009597